CLINICAL TRIAL: NCT06364982
Title: Distance Between Dental Implants as a Risk Indicator for Peri-implant Disease. A Multi-center Cross-sectional Study
Brief Title: Distance Between Dental Implants as a Risk Indicator for Peri-implant Disease.
Status: Recruiting | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Tiago Ribeiro Amaral, PhD candidate, Universitat Internacional de Catalunya
Other Study IDs: PER-ECL-2023-05
Record Dates: First submitted 2024-01-31; First posted 2024-04-15 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Peri-implant Mucositis; Peri-Implantitis
Keywords: Peri-implantitis; Peri-implant diseases; Peri-implant mucositis; Inter-implant distances
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inter-implant distance ≤ 3mm: Presence of an inter-implant distance ≤ 3mm
  Interventions: Diagnostic Test: Two contiguous dental implants placed with less ≤ 3mm from each other.
- Inter-implant distance ≥ 3mm: Presence of an inter-implant distance ≥ 3mm
  Interventions: Diagnostic Test: Two contiguous dental implants placed with > 3mm from each other.

INTERVENTIONS:
Diagnostic Test: Two contiguous dental implants placed with less ≤ 3mm from each other. — Implant Placement of 2 contiguous dental implants with less ≤ 3mm from each other.
  Groups: Inter-implant distance ≤ 3mm
Diagnostic Test: Two contiguous dental implants placed with > 3mm from each other. — Implant Placement of 2 contiguous dental implants with > 3mm from each other.
  Groups: Inter-implant distance ≥ 3mm

SUMMARY:
The aim of this study is to analyse contiguous dental implants and its peri-implant status depending on different inter-implant distances.

DETAILED DESCRIPTION:
The present research project has been designed as a multicentric cross-sectional study. The STROBE guidelines have been followed in the design of this observational study.

Ethical issues The study will be performed after the approval of the Ethics Committee of the Universitat Internacional de Catalunya (UIC) and Faculdade de Medicina Dentária da Universidade de Lisboa (FMDUL) and will be intended to be registered in clinicaltrials.gov. Also, this research will be conducted according to the principles outlined in the Declaration of Helsinki (revised, amended, and clarified in 2013). In addition, all study participants will provide written informed consent before participating in the study.

Study population Subjects will be selected from an electronic database collected at the CUO (UIC) / CU (FMDUL) and composed of patients treated with at least two contiguous dental implants before 2021. This investigation will use a stratified random sampling based on year of implant placement to select a representative sample of subjects with implant-supported restorations conducted during the period 2001-2020 at the CUO and CU. Then, two examiners (I.T. / F.F.) will contact patients by telephone once every 2 days (with a maximum of 3 attempts) for an evaluation by the same investigators (I.T / F.F).

Criteria for subject selection will be as follows:

* The patient must be ≥18 years of age and systemically healthy;
* Partially edentulous patients, rehabilitated until 2020 (i.e., a minimum of 3 years of function time) with at least two contiguous implant-supported restorations in the maxilla or mandible;
* Screw or cemented-retained prosthesis;
* Fixed dental prosthesis (i.e., single crowns and partial prosthesis);
* No implant mobility.

Moreover, the exclusion criteria will be the following:

* Pregnant and lactating women;
* Patients who have taken systemic antibiotics during the 3 months prior to the examination;
* Patients being treated with drugs that may induce a gingival overgrowth;
* Patients undergoing orthodontic treatment (since it can influence periodontal diagnosis);
* Patients who have received mechanical debridement during the 3 months prior to the exam;
* Patients who have received surgical treatment for peri-implantitis;
* Psychophysical inability to carry out study procedures.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be ≥18 years of age and systemically healthy;
* Partially edentulous patients, rehabilitated until 2020 (i.e., a minimum of 3 years of function time) with at least two contiguous implant-supported restorations in the maxilla or mandible;
* Screw or cemented-retained prosthesis;
* Fixed dental prosthesis (i.e., single crowns and partial prosthesis);
* No implant mobility.

Exclusion Criteria:

* Pregnant and lactating women;
* Patients who have taken systemic antibiotics during the 3 months prior to the examination;
* Patients being treated with drugs that may induce a gingival overgrowth;
* Patients undergoing orthodontic treatment (since it can influence periodontal diagnosis);
* Patients who have received mechanical debridement during the 3 months prior to the exam;
* Patients who have received surgical treatment for peri-implantitis;
* Psychophysical inability to carry out study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from an electronic database collected at the CUO (UIC) / CU (FMDUL) and composed of patients treated with at least two contiguous dental implants before 2021. This investigation will use a stratified random sampling based on year of implant placement to select a representative sample of subjects with implant-supported restorations conducted during the period 2001-2020 at the CUO and CU. Then, two examiners (I.T. / F.F.) will contact patients by telephone once every 2 days (with a maximum of 3 attempts) for an evaluation by the same investigators (I.T / F.F).
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of peri-implant diseases. | At least 36 months of function - at the moment of the evaluation
  Prevalence of peri-implant mucositis and peri-implantitis.

SECONDARY OUTCOMES:
FMPI | At least 36 months of function - at the moment of the evaluation
  Full Mouth Plaque Index
FMBI | At least 36 months of function - at the moment of the evaluation
  Full Mouth Bleeding Index
mPI | At least 36 months of function - at the moment of the evaluation
  modified Plaque Index
mBI | At least 36 months of function - at the moment of the evaluation
  modified Bleeding Index
SoP | At least 36 months of function - at the moment of the evaluation
  Suppuration on Probing
PPD | At least 36 months of function - at the moment of the evaluation
  Probing Pocket Depth
MR | At least 36 months of function - at the moment of the evaluation
  Mucosal Recession
KM | At least 36 months of function - at the moment of the evaluation
  Keratinized Mucosa
Implant location | At least 36 months of function - at the moment of the evaluation
  Implant location in the oral cavity
Implant position | At least 36 months of function - at the moment of the evaluation
  Implant position in the oral cavity
Implant type | At least 36 months of function - at the moment of the evaluation
  Implant type used
Implant brand | At least 36 months of function - at the moment of the evaluation
  Brand of the implant used
Implant roughness | At least 36 months of function - at the moment of the evaluation
  Type of implant roughness
Implant diameter | At least 36 months of function - at the moment of the evaluation
  Type of implant diameter
Implant length | At least 36 months of function - at the moment of the evaluation
  Length of the implant
Apico-coronal position of the implant | At least 36 months of function - at the moment of the evaluation
  Apico-coroal position
Inter-implant distances (IID) | At least 36 months of function - at the moment of the evaluation
  Inter-implant distance
Implant placement protocol | At least 36 months of function - at the moment of the evaluation
  Moment of the implant placement
Bone grafting procedures (BGP) at implant placement | At least 36 months of function - at the moment of the evaluation
  Bone grafting associated with the implant placement
Implant-supported restorations | At least 36 months of function - at the moment of the evaluation
  Screwed or Cemented
Cleansability of the prosthesis | At least 36 months of function - at the moment of the evaluation
  Cleansable, difficult or impossible to clean

CONTACTS AND LOCATIONS:
Overall Officials: Cristina V Vallès, PhD, Study Director — Department of Periodontology, University Internacional de Cataluña
Locations (1):
- Clínica Universitaria de Odontologia, Sant Cugat del Vallès, Barcelona, Spain

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT06364982/Prot_SAP_000.pdf